CLINICAL TRIAL: NCT02691650
Title: Point of Care Testing of Cholinesterase Activity During Burn- and Polytrauma
Acronym: POCCET
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Collaborators: BG Trauma Center Ludwigshafen (Other)
Responsible Party: Principal Investigator, Aleksandar Zivkovic, Dr. med. Aleksandar Zivkovic, University Hospital Heidelberg
Other Study IDs: Burns and Trauma POC ChE Study
Record Dates: First submitted 2016-02-16; First posted 2016-02-25 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Trauma; Burns
Keywords: serum cholinesterase; plasma cholinesterase; pseudocholinesterase; systemic inflammation; SIRS; polytrauma
MeSH Terms: conditions — Wounds and Injuries; Burns; Butyrylcholinesterase deficiency; Multiple Trauma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A miniature amount (10 μl) of whole blood is needed for the serum cholinesterase activity analysis. This blood specimen will be taken from otherwise routine blood gas analysis collection, taken upon arrival into the emergency room, as a part of the standardized ICU diagnostic and therapeutic procedure. The serum cholinesterase activity analysis, therefore, doesn't require additional blood collection.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- polytrauma patients: Patients with severe traumatic injury, admitted to the emergency unit. Serum cholinesterase activity measurement using 10 µl whole blood, otherwise obtained through routine blood gas analysis upon arrival to the hospital.
- burns patients: Patients with burns trauma, admitted to the emergency unit. Serum cholinesterase activity measurement using 10 µl whole blood, otherwise obtained through routine blood gas analysis upon arrival to the hospital.

SUMMARY:
Goal of this study is to measure serum cholinesterase activity in patients with traumatic and/or burns injury admitted to the emergency room by using point-of- care-test system (POCT). Serum cholinesterase activity, measured using POCT system, might play an important role in the early diagnosis and prediction of patient outcome in trauma-induced systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* signed written consent
* 18 years and older
* severe trauma (ISS > 15)
* burns injury (2. degree more than 15% body surface or 3 degree more than 10% body surface)
* SIRS

Exclusion Criteria:

* not fulfilling the inclusion criteria
* failure to adhere

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the emergency unit of the trauma and burns center
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2016-02; Primary Completion 2018-02 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Early diagnosis of the systemic inflammation by using the serum cholinesterase activity measurement | after completed patient recruitment, 1 year
  By using Point-of-care measurement of serum cholinesterase activity (U/l) and by observing a change in the enzyme activity over time (reduction of serum cholinesterase activity within the first 6 hours after traumatic injury) would allow an additional tool in early diagnosis and treatment of systemic inflammation.

SECONDARY OUTCOMES:
correlation of the cholinesterase activity and the trauma/disease severity scores | after completed patient recruitment, 1 year
  To evaluate the correlation of the serum cholinesterase activity change with the trauma severity, the obtained serum cholinesterase activities (U/l) will be compared to the trauma severity scores (ISS, %TBSA).

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Hofer, Prof. Dr., Principal Investigator — Department of Anesthesiology, Heidelberg University Hospital; Stefan Kleinschmidt, Prof. Dr., Study Chair — Department of Anaesthesia, Intensive Care Medicine and Pain Therapy, BG Trauma Centre Ludwigshafen, Ludwigshafen, Germany
Locations (1):
- Department of Anaesthesia, Intensive Care Medicine and Pain Therapy, BG Trauma Center Ludwigshafen, Ludwigshafen am Rhein, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No